CLINICAL TRIAL: NCT04593498
Title: Detection of Atrial Fibrillation in Patients With Excessive Supraventricular Activity
Brief Title: Excessive Supraventricular Activity and Atrial Fibrillation
Acronym: ESA-AF
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Johan Engdahl, MD, Associate Professor, Karolinska Institutet
Other Study IDs: ESA_AF2018
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Supraventricular Beat, Premature; Premature Supraventricular Beats; Premature Atrial Complex; Extrasystole, Atrial
Keywords: Excessive supraventricular ectopic activity
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Atrial Premature Complexes | interventions — Echocardiography; Caves; Blood Specimen Collection; Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 20 ml of plasma will be sampled at index and at 21 months in ESVEA and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESVEA: ESVEA (Excessive supraventricular ectopic activity): Participants with at least 30 supraventricular extra systole (SVES)/h or a supraventricular run of at least 20 beats.
  Interventions: Diagnostic Test: Holter recording; Diagnostic Test: Echocardiography (Echo); Diagnostic Test: Blood sample; Diagnostic Test: 24 hour ambulatory blood pressure monitoring And Arteriograph
- Non-ESVEA: Participants not meeting inclusion criteria
  Interventions: Diagnostic Test: Holter recording; Diagnostic Test: Echocardiography (Echo); Diagnostic Test: Blood sample; Diagnostic Test: 24 hour ambulatory blood pressure monitoring And Arteriograph

INTERVENTIONS:
Diagnostic Test: Holter recording — Holter recording with Zenicor Flex ECG during 14 days.
Diagnostic Test: Echocardiography (Echo) — Echocardiography: Comprehensive transthoracic echocardiography with special focus on atrial dimension and function.
Diagnostic Test: Blood sample — Blood sample: 2 x 10 ml EDTA plasma sampled from venous blood at index and at 21 months. Troponin T, NTproBNP, Na, K, Creatinine. Sample for Biobank for future analysis.
Diagnostic Test: 24 hour ambulatory blood pressure monitoring And Arteriograph — To assess artery stiffness.

SUMMARY:
The aim of the proposed study is to determine if individuals with excessive supraventricular ectopic activity (ESVEA) on Holter recording should be subjected to prolonged screening with Event loop recorder in order to detect previously undiagnosed Atrial fibrillation / flutter. Other biomarkers such as plasma biomarkers, high-end echocardiography and assessment of blood pressure and atrial stiffness will be studied and compared in ESVEA and control group as well as progression of atrial cardiomyopathy in ESVEA patients.

DETAILED DESCRIPTION:
Excessive supraventricular ectopic activities (ESVEA) are a common finding on long-term ECG recordings and have a connection to atrial cardiomyopathy, incident AF, stroke and mortality.

Holter recording from 2022 preformed at Danderyd hospital will be screened in order to identify 125 recordings with ESVEA, defined as at least 30 atrial ectopic beats/hour or a supraventricular run of at least 20 consecutive beats. Participants fulfilling eligibility criteria will be offered prolonged AF screening with continuous holter recording during 14 days. A matched control group (125 participants) without ESVEA will also be screened using same method.

Cardiovascular data from medical records will be collected in order to obtain information regarding co-morbidities and being able to assess CHA2DS2-VASC score. Participants will be asked to fill in a questionnaire.

Samples of blood will be collected at index time, after 21± 3 months for further analysis with the aim of identifying biomarkers for atrial fibrillation. During these two time periods echocardiography, 24 hour ambulatory blood pressure monitoring and assessment af artery stiffness with Arteriograph will also be preformed.

The study population will after 21± 3 months be subjected to renewed screening with Holter in order to examine the persistence of excessive supraventricular activity.

Four years after the completion of screening visits, data from patient records and information thorough telephone interview and/or data from Swedish Patient Register, Swedish Dispensed Drug Register will be collected

ELIGIBILITY:
Inclusion Criteria:

Patients with at least 30 supraventricular extra systole (SVES)/h or a supraventricular run of at least 20 beats on a Holter recording.

Exclusion Criteria:

Age < 70 years, >89 years Atrial fibrillation / flutter Lifelong treatment with oral anticoagulant Patients with implantable cardiac device Congestive heart failure (CHF) with Ejection fraction (EF) ≤ 30% Severe valvular heart disease

Ages: 70 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Individuals who have underwent Holter recording at Danderyd hospital after 2022.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
atrial fibrillation yield in extended ECG screening among patients with ESVEA on Holter recording as compared to patients without ESVEA. | 10-14 days
  Proportion of patients with at least one episode of atrial fibrillation with a duration of at least 30 seconds among patients with ESVEA on Holter recording as compared to patients without ESVEA.

SECONDARY OUTCOMES:
the clinical development of atrial fibrillation subtype in patients diagnosed with atrial fibrillation. | 2 years
  Presence of paroxysmal or permanent atrial fibrillation on follow-up.
Temporal development of ESVEA and atrial cardiomyopathy on repeated Holter recordings. | 2 years
  Comparison of burden of supraventricular extrasystolic beats and number of episodes and duration of longest episode of supraventricular tachycardia.
Temporal development of several blood biomarkers with a possible relation to atrial cardiomyopathy in patients with and without ESVEA. | 2 years
  Explorative sequential analysis of several blood biomarkers using PEA:
association between plasma biomarkers and the development of atrial fibrillation in patients with ESVEA. | 2 years
  Comparison of biomarker profile in patients diagnosed with atrial fibrillation and patients not diagnosed with atrial fibrillation.
Association between ESVEA, atrial fibrillation and other relevant comorbidities such as stroke, heart failure and major bleeding as well as mortality. | 4 years or longer
  Long-term data on incident stroke, heart failure, major bleedning and mortality compared between ESVEA- and non-ESVEA groups.
echocardiographic parameters in relation to ESVEA and/or AF. | 2 years
  Comparison of echocardiographic parameters with focus on atrial dimension and function compared between ESVEA and non-ESVEA group.
Artrial stiffness in relation to ESVEA and/or AF. | 2 yeras
  Comparison of artrial stiffness and blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No